CLINICAL TRIAL: NCT07314840
Title: Ultrasonographic Examination of Other Enthesitis Sites in Patients With Lateral Epicondylitis: A Cross-Sectional Study
Brief Title: Ultrasonographic Examination of Other Enthesitis Sites in Patients With Lateral Epicondylitis
Status: Recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, İlker Yağcı, Prof. M.D., Marmara University
Other Study IDs: 09.2025.25-0844
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Lateral Epicondylitis; Lateral Elbow Tendinopathy (Tennis Elbow)
Keywords: Lateral Epicondylitis; Lateral Elbow Tendinopathy; Tennis Elbow; Enthesitis; Madrid Sonographic Enthesitis Index; MASEI
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lateral Epicondylitis: Patients with lateral epicondylitis will be included in this group.
  Interventions: Diagnostic Test: Madrid Sonographic Enthesitis Index
- Control: Healthy volunteers with similar demographic characteristics will be enrolled to this group.
  Interventions: Diagnostic Test: Madrid Sonographic Enthesitis Index

INTERVENTIONS:
Diagnostic Test: Madrid Sonographic Enthesitis Index — Patients will be evaluated with ultrasound at 6 different locations on each side, for total of 12 locations. These will be insertion points of triceps brachii tendon, quadriceps tendon, proximal and distal patellar tendons, achilles tendon and the plantar fascia. Evaluation parameters are the structure and thickness of the tendon, the presence of calcifications or enthesophytes, erosions in the bone, regional bursitis, and the presence of power-Doppler signal in the entheses.
  Other Names: MASEI

SUMMARY:
Lateral epicondylitis (LE) is the tendinopathy of the common extensor tendon. Although exact etiology remains unclear, it is believed to be caused by overuse.

Even though, genetics factor related to tendinopathies were defined accompanying tendinopathies in patients with LE is yet to be studied.

Madrid sonographic enthesitis index (MASEI) is an ultrasound based scoring system, developed for the evaluation of the enthesitis. Initially developed for ankylosing spondylitis, its usage has also become widespread in other musculoskeletal diseases.

The aim of this study is to calculate the MASEI score in patients diagnosed with LE, and compare it to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Tenderness with palpation at the lateral epicondyle
* Pain aggravated with resisted wrist extension

Exclusion Criteria:

* History of rheumatologic diseases
* History of elbow, knee or ankle surgery
* History of corticosteroid injections on elbow, knee or ankle
* History of peripheral neuropathy
* Acute trauma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients presented to the outpatient clinic of Physical Medicine and Rehabilitation of Marmara University with elbow pain and diagnosed with lateral epicondylitis will be informed about the study. Willing patients will be enrolled after written consent is taken.
  Control group will be chosen with volunteers, which have similar demographic characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Madrid Sonographic Enthesitis Index | At enrollment
  Patients will be evaluated with ultrasound at 6 different locations on each side, for total of 12 locations. At each location; structure and thickness of the tendon, the presence of calcifications or enthesophytes, erosions in the bone, regional bursitis, and the presence of power-Doppler signal will be noted. Each parameter has a point of its own. Points obtained from each parameter will be added and total MASEI score (0-136) will be calculated. Higher scores indicate the presence of enthesitis.

CONTACTS AND LOCATIONS:
Overall Officials: İlker Yağcı, Prof. Dr., Principal Investigator — Acıbadem Ataşehir Hospital
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to legal restrictions, all data will be anonymized. Individual participant data won't be shared to third parties.

REFERENCES:
- [Background] Ozsoy-Unubol T, Yagci I. Is ultrasonographic enthesitis evaluation helpful for diagnosis of non-radiographic axial spondyloarthritis? Rheumatol Int. 2018 Nov;38(11):2053-2061. doi: 10.1007/s00296-018-4164-4. Epub 2018 Oct 9. PMID 30302556
- [Background] de Miguel E, Cobo T, Munoz-Fernandez S, Naredo E, Uson J, Acebes JC, Andreu JL, Martin-Mola E. Validity of enthesis ultrasound assessment in spondyloarthropathy. Ann Rheum Dis. 2009 Feb;68(2):169-74. doi: 10.1136/ard.2007.084251. Epub 2008 Apr 7. PMID 18390909
- [Background] Okur SC, Dogan YP, Mert M, Aksu O, Burnaz O, Caglar NS. Ultrasonographic Evaluation of Lower Extremity Entheseal Sites in Diabetic Patients Using Glasgow Ultrasound Enthesitis Scoring System Score. J Med Ultrasound. 2017 Jul-Sep;25(3):150-156. doi: 10.1016/j.jmu.2017.03.011. Epub 2017 May 6. PMID 30065480
- [Background] Johns N, Shridhar V. Lateral epicondylitis: Current concepts. Aust J Gen Pract. 2020 Nov;49(11):707-709. doi: 10.31128/AJGP-07-20-5519. PMID 33123709
- [Background] Karanasios S, Korakakis V, Moutzouri M, Drakonaki E, Koci K, Pantazopoulou V, Tsepis E, Gioftsos G. Diagnostic accuracy of examination tests for lateral elbow tendinopathy (LET) - A systematic review. J Hand Ther. 2022 Oct-Dec;35(4):541-551. doi: 10.1016/j.jht.2021.02.002. Epub 2021 Feb 27. PMID 33814224